CLINICAL TRIAL: NCT01722981
Title: Percutaneous Tracheostomy - Systematic Comparison Among Three Methods: US-guided Tracheostomy, Bronchoscopy Guided Tracheostomy, and Direct Laryngoscopy Tracheostomy.
Brief Title: Percutaneous Tracheostomy - Systematic Comparison Among Three Methods: Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TASMC-12-PS-0408-12-CTIL
Record Dates: First submitted 2012-11-04; First posted 2012-11-07 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Other Tracheostomy Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Direct laryngoscopy (Active Comparator): Performing percutaneous tracheostomy as accepted in our institute: By placing the tube higher up near the vocal cords by direct laryngoscopy. In the second stage tracheal perforation by a needle will be carried out by palpation of the anatomical placement of the neck.
  Interventions: Procedure: Percutaneous tracheostomy
- Real time sonography (Active Comparator): Percutaneous tracheostomy will be guided by real time sonography (with the visualization of the needle path) using acoustic shadows of the cricoid and the tracheal rings.
  In both methods, in order to identify the anatomic location of the needle prick- after passing the guide wire, the front elevation will be verified by optical means, which will be drawn out immediately afterwards.
  Interventions: Procedure: Percutaneous tracheostomy
- Bronchoscopy (Active Comparator): Percutaneous tracheostomy will be guided by bronchoscopy. Initially, the tube will be placed according to the desired height observed by the bronchoscope, phase two will be tracheal perforation by a needle under trans illumination and real-time view on the income of the needle and the passage of the guide wire.
  Interventions: Procedure: Percutaneous tracheostomy

INTERVENTIONS:
Procedure: Percutaneous tracheostomy — Three methods of percutaneous tracheostomy

SUMMARY:
Percutaneous tracheostomy is routinely performed in most intensive care units in the world.Several studies have shown that the procedure is safe and economically efficient in comparison to open surgical operation in the operating room.

In our institution as in a number of institutions in the country, it is acceptable to perform the operation by placing the tube on a high position near the vocal cords by direct laryngoscopy and then puncturing the trachea with a needle, by location of the anatomy by palpation of the neck.

Using technological aids, such as direct sonography and bronchoscopy in real time may significantly reduce the rate of complications as a result of performing percutaneous tracheostomy.

So far, no systematic comparison has been made among the three methods.

DETAILED DESCRIPTION:
Percutaneous tracheostomy is routinely performed in most intensive care units in the world in a number of indications, such as: airway obstruction, need for a long respiratory support, improvement in respiratory toilet, prophylaxis before head and neck procedures and cases of severe obstructive sleep apnea.

Several studies have shown that the procedure is safe and economically efficient in comparison to open surgical operation in the operating room.

In many places around the world it is customary in to perform the operation under the guidance of a bronchoscope to prevent damage to adjacent structures, high or low position of the tube, and damage to the posterior wall of the trachea and to approve the final position of the tube. However, the use of a bronchoscope depends on the availability of the equipment, knowledge of the operator, temporary occlusion of the trachea and hypercarbia, increased length of the procedure, and maintenance cost (disinfection, replacement, etc.).

Ultrasound that is performed before percutaneous procedure may be useful in preventing damage to para tracheal adjacent structures, and preventing high placement of the tube. The use of duplex sonography with real-time visualization of the needle path is done routinely in procedures such as central venous catheterization, and may improve the safety and accuracy of percutaneous tracheostomy without causing airway obstruction or hypercarbia. Feasibility of the procedure has been reviewed in an article by Rajajee et al .

In our institution as in a number of institutions in the country, it is acceptable to perform the operation by placing the tube on a high position near the vocal cords by direct laryngoscopy and then puncturing the trachea with a needle, by location of the anatomy by palpation of the neck.

So far, no systematic comparison has been made among the three methods.

ELIGIBILITY:
Inclusion Criteria:

* All intubated patients with various injuries requiring percutaneous tracheostomy (in- house and out- house patients)
* Minimal age 18

Exclusion Criteria:

* No patient consent for participation.
* Anatomical problem which does not allow for percutaneous tracheostomy and requires open procedure in the operating room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Systematic comparison | 3 years
  a systematic comparison among the three methods of percutaneous tracheostomy in terms of safety: minor and major periprocedural morbidity and mortality, up to 30 days.

SECONDARY OUTCOMES:
Minor morbidity | 3 years
  Minor morbidity among patients, and a comparison between the in-house patients to the rest of hospitalized patients that come to the unit for the procedure, according to the same criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sorkine, professor, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel